CLINICAL TRIAL: NCT03683680
Title: Prospectively Collected Pleural Biopsies for Validation of Malignant Pleural Mesothelioma Prognostic Biomarkers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Raphael Bueno, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-220; CA120528 (Other: NCI)
Record Dates: First submitted 2018-09-21; First posted 2018-09-25 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-02

CONDITIONS: Mesothelioma
Keywords: Mesothelioma
MeSH Terms: conditions — Mesothelioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRiS (Experimental): * The specimens to be collected will include at least five pleural biopsy samples
  * MPT test and the CLDN15/VIM test will be performed
  Interventions: Other: MPT Test; Other: CLDN15/VIM Test

INTERVENTIONS:
Other: MPT Test — molecular expression tests at the RNA level using approximately 7 or more genes with RTPCR, nanostring or similar platforms
Other: CLDN15/VIM Test — molecular expression tests at the RNA level using approximately 7 or more genes with RTPCR, nanostring or similar platforms

SUMMARY:
This research study is evaluating a new method for determining stage and prognosis of individuals with malignant pleural mesothelioma.

DETAILED DESCRIPTION:
The purpose of this research study is to test a new method for determining the stage and prognosis of patients with malignant pleural mesothelioma. Currently, it is not possible to accurately determine cancer stage prior to surgery or another treatment. This new method may allow doctors to better classify cancer stage and give a better estimate for prognosis prior to surgery or another treatment.

In this research study, the investigators would like to use biopsied tissue to study certain characteristics that will help test the new method for determining cancer stage and estimating prognosis.

In this research study, the investigators are...

* Obtaining pleural specimens at the time of routine diagnostic biopsy during the participant's standard treatment.
* Storing your biopsied tissue
* Studying the tissue to determine if the new method of staging and prognosis is accurate and valid

ELIGIBILITY:
Inclusion Criteria:

* All adult patients with a diagnosis of malignant pleural mesothelioma undergoing

  * diagnostic pleural biopsy
  * pleuroscopy
  * and/or VATS resections
* Participants must be 18 years of age or older.

Exclusion Criteria:

-Any patient who is found to be unsuitable for

* surgery,
* treatment
* diagnosis,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2018-10-31 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-10-01 (Estimated)

PRIMARY OUTCOMES:
Pre-treatment Prognostic Algorithm Validation | 4 years
  The primary objective is to utilize a novel prognostic algorithm to predict the outcome of MPM patients. This algorithm includes 4 different tests: molecular, radiological, and blood based. It will be performed on 240 prospectively-collected samples. A score of 0-4 will be assigned to each patient and the data will be analyzed by a statistician

SECONDARY OUTCOMES:
Evaluation of Molecular Tests Base on RNA Expression | 4 years
  The secondary objective is to develop new molecular signatures for distinct clusters of mesothelioma samples grouped according to their gene expression. RNA expression data will be compared between one cluster and all the other clusters and using a variety of statistical and bioinformatics tools. Two-hundred sixteen MPM cases with available RNAseq data will be divided into training and test sets to develop and test potential signatures. The signatures that define each cluster with high sensitivity and specificity will then be tested using RTPCR in a cohort of 555 prospective-collected samples.

CONTACTS AND LOCATIONS:
Overall Officials: Raphael Bueno, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No